CLINICAL TRIAL: NCT04551950
Title: Safety Study of Bintrafusp Alfa in Combination With Other Anti-cancer Therapies in Participants With Locally Advanced or Advanced Cervical Cancer (INTR@PID 046)
Brief Title: Bintrafusp Alfa Combination Therapy in Participants With Cervical Cancer (INTR@PID 046)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0046; 2020-001561-36 (EudraCT Number)
Record Dates: First submitted 2020-09-07; First posted 2020-09-16 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer
Keywords: Advanced cervical cancer; Bintrafusp alfa; M7824; INTR@PID; Transforming growth factor-beta; Programmed death-ligand 1
MeSH Terms: conditions — Uterine Cervical Neoplasms; Camurati-Engelmann Syndrome | interventions — bintrafusp alfa protein, human; Carboplatin; Paclitaxel; Bevacizumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1A:M7824+Cisplatin/Carboplatin+Paclitaxel+Bevacizumab (Experimental)
  Interventions: Drug: M7824; Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab; Drug: Cisplatin
- Cohort1B:M7824+Cisplatin or Carboplatin+Paclitaxel (Experimental)
  Interventions: Drug: M7824; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin
- Cohort 2: M7824+Cisplatin+ Radiotherapy (Experimental)
  Interventions: Drug: M7824; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: M7824 — Participants received bintrafusp alfa until confirmed disease progression, death, unacceptable toxicity and study withdrawal maximum of 2 years (at the discretion of the Investigator).
  Other Names: Bintrafusp alfa
Drug: Carboplatin — Carboplatin was administered intravenously as per standard of care.
  Arms: Cohort 1A:M7824+Cisplatin/Carboplatin+Paclitaxel+Bevacizumab; Cohort1B:M7824+Cisplatin or Carboplatin+Paclitaxel
Drug: Paclitaxel — Paclitaxel was administered intravenously as per standard of care.
  Arms: Cohort 1A:M7824+Cisplatin/Carboplatin+Paclitaxel+Bevacizumab; Cohort1B:M7824+Cisplatin or Carboplatin+Paclitaxel
Drug: Bevacizumab — Bevacizumab was administrated as indicated for standard of care.
  Arms: Cohort 1A:M7824+Cisplatin/Carboplatin+Paclitaxel+Bevacizumab
Drug: Cisplatin — Cisplatin was administered intravenously as per standard of care.
Radiation: Radiotherapy — Participants received radiotherapy as per standard of care.
  Arms: Cohort 2: M7824+Cisplatin+ Radiotherapy

SUMMARY:
This study was to evaluate the safety and tolerability of bintrafusp alfa in combination with other anti-cancer therapies in participants with locally advanced or advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for participants enrolling into Cohort 1:
* Study participants had documented persistent, recurrent, or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix
* Study participants had not been treated with systemic chemotherapy and were not amenable to curative treatment
* Prior radiation with or without radio-sensitizing chemotherapy was allowed
* Inclusion Criteria for participants enrolling into Cohort 2:
* Participants had documented evidence of cervical adenocarcinoma, squamous cell carcinoma, or adenosquamous carcinoma International Federation of Gynecology and Obstetrics (FIGO) 2018 Stages 1B2 to 4A
* Participants had not received prior chemotherapy or radiotherapy for cervical cancer
* Inclusion Criteria for all participants:
* Archival tumor tissue sample or newly obtained core or excisional biopsy was required
* Participants who had Eastern Cooperative Oncology Group (ECOG) Performance status (PS) of 0 to 1 were eligible
* Participants had a life expectancy greater than or equal to 12 weeks
* Participants had adequate hematological, hepatic, renal, and coagulation function as defined in the protocol
* Participants with known Human immunodeficiency virus (HIV) infections were eligible if the criteria described in the protocol were met
* Participants with Hepatitis B virus (HBV) and/or Hepatitis C virus (HCV) infections were eligible if the criteria described in the protocol were met
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Exclusion Criteria for All Participants were:
* Participants with active central nervous system (CNS) metastases causing clinical symptoms or metastases that required therapeutic intervention were excluded. Participants with a history of treated CNS metastases (by surgery or radiation therapy) were not eligible unless they had fully recovered from treatment, demonstrated no progression for at least 4 weeks, and were not using steroids for at least 7 days prior to the start of study intervention
* Participants that received any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that did not require immuno-suppression
* Participants with significant acute or chronic infections
* Participants with active autoimmune disease that might have deteriorated when receiving an immuno-stimulatory agent
* Participants with clinically significant cardiovascular/cerebrovascular disease including: a cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure, or serious cardiac arrhythmia
* Participants with a history of bleeding diathesis or recent major bleeding events
* Participant that had received prior cancer treatment with any other immunotherapy or checkpoint inhibitors or any other immune-modulating monoclonal antibody (mAb)
* Exclusion Criteria for Participants in Cohort 1A related to use of bevacizumab were:
* Participants with inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Participants with significant vascular disease within 6 months prior to Screening
* Participants with a history of hemoptysis within 1 month prior to Screening
* Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
* Participants with a history of abdominal or trache-oesophageal fistula or gastrointestinal (GI) perforation within 6 months prior to Screening
* Participants with clinical signs of GI obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Participants with evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Participants with serious, non-healing wound, active ulcer, or untreated bone fracture
* Participants with proteinuria
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (13):
- United States (5):
  - Stanford Health Care Hospital & Clinics, Stanford, California
  - Augusta University - formerly Georgia Regents University, Augusta, Georgia
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - University of Cincinnati Physicians Group, LLC - Pharmatech Oncology, Inc, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
- Japan (5):
  - National Cancer Center Hospital, Chūōku
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Sunto-gun
- Spain (3):
  - Hospital Clinic i Provincial de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, Barcelona

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0046
- See also: US Medical Information website, Medical Resources — http://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 participants were screened out of which 25 participants were treated.
Groups:
- Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab: Participants received 2400 miligrams (mg) Bintrafusp alfa along with 50 milligram per square meter (mg/m^2) Cisplatin or Carboplatin, Paclitaxel and 15 milligram per kilogram (mg/kg) Bevacizumab every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
- Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel: Participants received 2400 mg Bintrafusp alfa along with 50 mg/m^2 Cisplatin or Carboplatin, 175 mg/m^2 Paclitaxel every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
- Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy: Participants received 2400 mg Bintrafusp alfa once every 3 weeks along with 40 mg/m^2 Cisplatin weekly for 5 weeks followed by radiotherapy as per standard care.
Period: Overall Study
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Started | 8 | 9 | 8
Treated | 8 | 9 | 8
Completed | 8 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy | Total
Number analyzed (Participants) | 8 | 9 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (9) | 47 (8.3) | 49 (13.1) | 47 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 8 | 25
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 4 | 6 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Missing | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 9 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as Adverse Events (AEs) with any of following toxicities: Grade 4 nonhematologic toxicity or hematologic toxicity lasting more than equal to (>=) 7 days despite medical intervention; Grade 3 nausea, vomiting, and diarrhea lasting >= 3 days despite supportive care; Any Grade 3 or Grade 4 nonhematologic lab value leading to hospitalization or persisting for >= 7 days; Grade 3 or Grade 4: grade 3 is defined as absolute neutrophil count (ANC) less than (<) 1,000/mm3 with a temperature of > 38.3 degree Celsius (°C); grade 4 is defined as ANC < 1,000/mm3 with a temperature of > 38.3°C, with life-threatening consequences; Thrombocytopenia < 25,000/mm3 associated with bleeding not resulting in hemodynamic instability or a life-threatening bleeding resulting in urgent intervention; Bleeding events >= Grade 3 occurring within 5 days of bintrafusp alfa treatment; Prolonged delay (> 3 weeks) in initiating Cycle 2 due to treatment-related toxicity; Grade 5 toxicity.
Time Frame: Up to 4 weeks after first administration of study intervention
Population: Dose-Limiting Toxicity Analysis (DLT) Set included all participants who completed the DLT period (within 4 weeks after first administration of study intervention) with at least 80 Percent (%) of the planned cumulative dose received during this period for each study intervention and/or who experienced at least one DLT during the DLT period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 8 | 9 | 8
Participants | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Treatment-Emergent Adverse Events (TEAEs) were defined as events with onset date or worsening during the on-treatment period. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs included serious TEAEs and non-serious TEAEs.
Time Frame: Time from first treatment assessed up to approximately 20 months
Population: The safety (SAF) analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 8 | 9 | 8
Participants
  Any TEAEs | 8 | 9 | 8
  Any Serious TEAEs | 7 | 4 | 6

3. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of Bintrafusp Alfa
Description: Ceoi was the observed concentration at the end of the infusion period. This was taken directly from the observed Bintrafusp Alfa concentration-time data.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Serum Trough Concentration Levels (Ctrough) of Bintrafusp Alfa
Description: Ctrough was the serum concentration observed immediately before next dosing.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Bintrafusp Alfa
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Bintrafusp Alfa
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Bintrafusp Alfa
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Bintrafusp Alfa
Description: The time to reach the maximum observed concentration collected during a dosing interval. Tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Bintrafusp Alfa
Description: Elimination Half Life (T1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. Elimination half-life determined as 0.693/ Lamda z(λz), λz=terminal first order (elimination) rate constant.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of Bintrafusp Alfa
Description: A validated method was applied to detect ADAs in the presence of drug in human serum. The ADA titers of positive samples were determined.
Time Frame: Pre-dose Up to 20 months
Population: As per changes in planned analysis, the outcome measure related to immunogenicity were not assessed.
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Japanese Participants With Dose-Limiting Toxicities (DLTs)
Description: as for outcome 1
Time Frame: Up to 4 weeks after first administration of study intervention
Population: Dose-Limiting Toxicity Analysis (DLT) Set included all participants who completed the DLT period (within 4 weeks after first administration of study intervention) with at least 80 Percent (%) of the planned cumulative dose received during this period for each study intervention and/or who experienced at least one DLT during the DLT period. Number of Participants Analyzed=participants evaluable for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 2 | 0

12. Secondary Outcome: Number of Japanese Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Treatment-Emergent Adverse Events (TEAEs) were defined as events with onset date or worsening during the on-treatment period. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Time Frame: Time from first treatment assessed up to approximately 20 months
Population: The safety (SAF) analysis set included all participants who were administered any dose of any study intervention. Number of Participants Analyzed=participants evaluable for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Any TEAEs | 3 | 3 | 3
  Any Serious TEAEs | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: Time from first treatment assessed up to approximately 20 months
Arm/Group | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy
All-Cause Mortality (participants affected / at risk) | 2/8 | 2/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 7/8 | 4/9 | 6/8
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab (N=8) | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel (N=9) | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Uterine abscess (Infections and infestations) | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: Bintrafusp Alfa +Cisplatin/Carboplatin+Paclitaxel+Bevacizumab (N=8) | Cohort1B: Bintrafusp Alfa +Cisplatin or Carboplatin+Paclitaxel (N=9) | Cohort 2: Bintrafusp Alfa + Cisplatin+ Radiotherapy (N=8)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 3 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 6
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 4
Asthenia (General disorders) | 3 | 2 | 2
Catheter site pain (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 2 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 (0) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 1
Uterine abscess (Infections and infestations) | 1 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0
Amylase increased (Investigations) | 1 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 3 | 2 | 1
Lymphocyte count decreased (Investigations) | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 2
Platelet count decreased (Investigations) | 2 | 3 | 2
Weight decreased (Investigations) | 0 | 1 | 2
White blood cell count decreased (Investigations) | 2 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1 | 3
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 2 | 4 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Thrombosis in device (Product Issues) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Menopause (Social circumstances) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT04551950/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04551950/SAP_001.pdf